CLINICAL TRIAL: NCT07256119
Title: Evaluation of the Effect of Alpha Lipoic Acid on Radiation Induced Dermatitis in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana mohamed, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHDIRB2020110301 REC # 283
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Prevention
Keywords: Radiation Induced Dermatitis; RID; Alpha Lipoic Acid; Breast Cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- alpha lipoic acid (Experimental): patients will receive alpha lipoic acid 300 mg three times daily under the trade name of THIOTACID manufactured by EVAPHARMA for prophylaxis of the radiation-induced dermatitis (RID) from day 1 of radiation therapy till the end of the study.
  Interventions: Dietary Supplement: Alpha Lipoic Acid
- Control (No Intervention): patients will not receive any prophylactic intervention as there is no standard of care for prophylaxis to the radiation-induced dermatitis (RID).

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid — alpha lipoic acid 300 mg three times daily under the trade name of THIOTACID manufactured by EVAPHARMA.
  Arms: alpha lipoic acid

SUMMARY:
the purpose of this study is to evaluate the Effect of Alpha Lipoic Acid on Radiation Induced Dermatitis in Breast Cancer Patients

DETAILED DESCRIPTION:
Cancer is one of the leading causes of mortality worldwide, and cancer treatment options include chemotherapy, radiotherapy, surgery, and hormone therapy. Radiation therapy is a treatment based on the use of high-energy waves or radioactive particles to damage tumor cells to attenuate their growth. This modality has been effectively used for cancer treatment in more than 100 years.

Radiation therapy (RT) is one of the standard protocols with a high success rate for the treatment of breast cancer to reduce the risk of recurrence and death. The goal of radiation therapy is to destroy tumor cells with minimal damage to normal tissue. However, normal cells may be damaged when exposed to radiation.

Radiation-induced dermatitis (RID) occurs in 95% of patients receiving radiation therapy during their treatment. The skin cells located in close vicinity to the tumor cells receive large amounts of radiation, causing several complications such as redness, dry and wet desquamation, and tissue necrosis.

The occurrence of these complications in patients leads to discomfort, limited daily activities, and even stops radiotherapy, which negatively affects the cancer treatment. Symptoms usually appear 10-14 days following the initiation of treatment and carry on for 2 to 4 weeks during radiation therapy. Previous studies evaluated the effect of various topical and oral formulations in radiation-induced dermatitis. However, until now, there is no standard measure for the prevention of radiation-induced dermatitis in patients with breast cancer.

The mechanisms associated with radiation-induced dermatitis include inflammatory response and oxidative stress (OS). Inflammatory response and oxidative stress interact and promote each other. After radiation-induced cell damage, cells die in various forms, especially mitotic death, leading to inflammation and chronic oxidative stress. Understanding the mechanisms of chronic oxidative damage and injury of affected cells, tissues, and organs after exposure to radiation therapy may contribute to the development of treatment and management strategies of the complications associated with radiation therapy.

Inflammatory response

In the initial period of radiation therapy, there is an immediate generation of an inflammatory response. The early inflammatory response to radiation is mainly caused by pro-inflammatory cytokines (IL-1, IL-3, IL-5, IL-6, and tumor necrosis factor [TNF]-a), chemokines (eotaxin and IL-8), receptor tyrosine kinase, and adhesions molecules (intercellular adhesion molecule 1 [ICAM-1], E-selectin, and vascular cell adhesion protein). These factors can create a local inflammatory response of eosinophils and neutrophils, leading to self-perpetuating tissue damage and loss of protective barriers.

Oxidative stress (OS)

Chronic oxidative stress participates in the development of several diseases. The redox system plays a key role in the early and late effects of radiation-induced skin reactions (RISRs).

As 80% of the tissues and cells are made of water, much of the radiation damage from exposure to low linear energy transfer radiation (Photon& electrons) is due to radiolysis of water leading to the generation of reactive oxygen species (ROS) and reactive nitrogen species (RNS), which are important mediators for some cellular processes such as immune response, cell signaling, microbial defenses, differentiation, cell adhesion, and apoptosis. The reactive oxygen species and reactive nitrogen species are the major sources of normal tissue damage after exposure to radiation therapy. The production of reactive oxygen species undergoes molecular changes, damaging DNA, lipids, and proteins and activating early-response transcription factors and signal transduction pathways. As a result, it causes damage to the skin tissue.

Inflammation plays a key role in redox activation. Direct exposure of normal cells to IR or ROS leads to nuclear and mitochondrial DNA damage, which may result in cell death through apoptosis and necrosis. Cell apoptosis can trigger the release of anti-inflammatory cytokines such as interleukin-10 (IL-10) and Transforming Growth Factor-beta (TGF-β), while necrosis may cause the release of pro-inflammatory cytokines such as interleukin-1 (IL-1), interleukin-6 (IL-6),interleukin-8 (IL-8),interleukin-13 (IL-13), interleukin-33 (IL-33), and tumor necrosis factor alpha (TNF-a) and other inflammatory mediators.

It is known that oxygen radicals and nitrogen-centered radicals regulate transcription factors, such as nuclear factor kappa-light-chain-enhancer of activated B cells (NF-KB) and activator protein 1 (AP-1). NF-KB can be activated by cellular exposure to ultraviolet or ionizing radiation, infection, or trauma. This stimulus results in the dissociation of the inhibitory portion of the molecule, followed by translocation of NF-KB to the nucleus; the result in expression of genes that are linked to the inflammatory response.

Based on literature, Alpha-lipoic acid (ALA) is a pleiotropic medication with anti-inflammatory and antioxidant properties, of which the effects are exerted through the modulation of NF-kB which modulates inflammatory cytokines, including interleukin -1β (IL-1β) and interleukin-6 (IL-6), in different cell types and tissues. Additionally, Alpha-lipoic acid has the ability to combat oxidative damage via quenching a variety of intracellular free radicals. In addition, alpha-lipoic acid is involved in the recycling of some other natural cellular reactive oxygen species scavengers such as ascorbic acid, α-tocopherol, and glutathione (GSH).

Hence, many clinical trials have been using Alpha Lipoic Acid, to see its anti-inflammatory and antioxidant effects in different indications including Alzheimer's disease patients as Studies recently showed that interleukin -1β (IL-1β) and interleukin-6 (IL-6) DNA methylation is modulated in the brain of Alzheimer's disease patients. and alpha-lipoic acid induced repression of interleukin -1β (IL-1β) and interleukin-6 (IL-6) was dependent on DNA methylation, several studies show that alpha-lipoic acid has greet effect on patients with metabolic syndrome as it diminishes pro-inflammatory markers and enhances endothelial function, elements that are indicated in the pathogenesis of atherosclerosis. Along with that, it was also found that alpha-lipoic acid supplementation improved serum adiponectin and interleukin-6 (IL-6) levels, without changing serum liver enzymes and liver steatosis in obese patients with Non-alcoholic fatty liver disease, and in Diabetic patients with neuropathy treated with alpha-lipoic acid 600 mg daily for three weeks, have reduced pain, paresthesia, and numbness.

Previous studies demonstrated the safety and tolerability of alpha-lipoic acid in doses ranging from 600-1800 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years.
* Histologically confirmed invasive, early-stage breast carcinoma scheduled for adjuvant radiotherapy.
* Receiving total radiation dose of 40 Gy for 15 sessions.

Exclusion Criteria:

* Prior exposure to radiotherapy.
* Inflammatory or metastatic breast carcinoma.
* Patients with connective tissue disorders.
* Patients with skin inflammatory diseases (e.g. ectopic dermatitis).
* Patients with known allergy or hypersensitivity to alpha lipoic acid.
* Concomitant use of nonsteroidal anti-inflammatory drugs, corticosteroids, or antioxidant medications.
* Patients who will fail to sign the written consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of development of radiation induced dermatitis (RID) | weekly after every fifth Radiotherapy session till the end of study (3 weeks).
  If the patient developed Radiation induced dermatitis or not.
Evaluation of the Severity of radiation-induced dermatitis (RID) developed | weekly after every fifth Radiotherapy session till the end of study (3 weeks).
  severity will be scored using the Radiation Therapy Oncology Group (RTOG) criteria based on the clinical presentation.
Evaluation of Inflammatory biomarker level (Interleukin-6) | baseline, end of study Up to 3 Weeks
  Assessing Serum level of Interleukin-6 (IL6) using ELISA kits.
Evaluation of Incidence of Treatment-Emergent Adverse Events | weekly after every fifth Radiotherapy session till the end of study (3 weeks).
  Patients will be educated and instructed to report any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Mohamed Elsayed Kelany Abdelkader, Principal Investigator — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt